CLINICAL TRIAL: NCT06426355
Title: The Effeciency of Nicotinamide Mononucleotide (NMN) in Improving IVF/ICSI-ET Pregnancy Outcomes in Patients With Decreased Ovarian Reserve（DOR): a Randomized Double-blind Placebo Control Clinical Trail
Brief Title: The Effeciency of NMN in Improving IVF/ICSI-ET Pregnancy Outcomes in Patients With DOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M2023557
Record Dates: First submitted 2024-03-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Diminished Ovarian Reserve

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMN intervention (Active Comparator): Dietary Supplement: NMN intervention NMN capsules (total of 600mg/day) for 2-5 months
  Interventions: Dietary Supplement: NMN
- Placebo intervention (Placebo Comparator): Placebo NMN-free placebo capsules for 2-5 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NMN — NMN capsules (total of 600mg/day) for 2-5 months
  Arms: NMN intervention
Other: Placebo — NMN-free placebo capsules for 2-5 months
  Arms: Placebo intervention

SUMMARY:
The purpose of the study is to understand the effect of nicotinamide mononucleotide (NMN) on patients with diminished ovarian reserve and the outcomes of IVF/ICSI-ET.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are 20 to 40 years old.
2. At least two of the following three conditions should be met:

   1. The concentrations of anti-Mullerian hormone < 1.1 ng/ml,
   2. the values of antral follicle count was less than 7
   3. serum concentrations of day-3 follicle-stimulating hormone (FSH)： 10 IU/L ≤ FSH<20 IU/L
3. Individuals who can insist on continuous monitoring in the outpatient clinic.
4. Individuals who are not participating in other research projects currently or 3 months before the intervention.

Exclusion Criteria:

1. Individuals who are during pregnant, lactation or menopause.
2. Individuals who had non-46-XX karyotype, or attributed to known genetic etiology.

   Individuals who had pelvic surgery.
3. Cancer patients or receiving chemo/radiotherapy treatment within the past 5 years.
4. Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
5. Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.
6. Use of medications or traditional Chinese medicine that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 3 months.
7. Individuals who take niacin, nicotinamide, or other vitamin B3-related supplementation, or other supplementation such as coenzyme Q10, vitamin E currently or within the past 3 months.
8. Use of antibiotics, probiotics, or prebiotics that affect the flora within the past 3 months.
9. Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.
10. A medical history of severe cardiovascular and cerebrovascular diseases.
11. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.
12. Individuals who drink more than 15g of alcohol per day or have a smoking habit.
13. Individuals who need drug treatment for any mental illness such as epilepsy and depression.
14. Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.
15. Unable or unwilling to follow the study protocol.

Individuals who are during pregnant, lactation or menopause. Individuals who had non-46-XX karyotype, or attributed to known genetic etiology.

Individuals who had pelvic surgery. Cancer patients or receiving chemo/radiotherapy treatment within the past 5 years.

Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.

Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.

Use of medications or traditional Chinese medicine that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 3 months.

Individuals who take niacin, nicotinamide, or other vitamin B3-related supplementation, or other supplementation such as coenzyme Q10, vitamin E currently or within the past 3 months.

Use of antibiotics, probiotics, or prebiotics that affect the flora within the past 3 months.

Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.

A medical history of severe cardiovascular and cerebrovascular diseases. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.

Individuals who drink more than 15g of alcohol per day or have a smoking habit. Individuals who need drug treatment for any mental illness such as epilepsy and depression.

Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.

Unable or unwilling to follow the study protocol.

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The clinical pregnancy rate | through study completion, an average of 2 year
  The pregnancy rate of IVF/ICSI-ET

SECONDARY OUTCOMES:
Endocrine hormones including AMH | Within three months after the end of treatment with NMN or placebo
  Changes in endocrine hormones including AMH levels in serum after the intervention.
Follicle number | Within three months after the end of treatment with NMN or placebo
  The number of all antral follicles in each ovary will be determined using transvaginal ultrasonography for each participant.
In vitro fertilization - outcome indicators of embryo culture | Day of oocyte retrieval and 1 week after oocyte retrieval。Within three months after the end of treatment with NMN or placebo
  Number of oocytes obtained, number of MII oocytes, fertilization rate, number of available embryos, number of high-quality embryos, cycle cancellation rate
Biochemical pregnancy rate | after pregnancy and infant borned. Within 1 year after the end of treatment with NMN or placebo
  Biochemical pregnancy rate
live birth rate | after pregnancy and infant borned.Within 1 year after the end of treatment with NMN or placebo
  live birth rate
abortion rate | after pregnancy and infant borned.Within 1 year after the end of treatment with NMN or placebo
  abortion rate
pregnancy complications | after pregnancy and infant borned.Within 1 year after the end of treatment with NMN or placebo
  pregnancy complications, the condition of newborn births
the condition of newborn births | after pregnancy and infant borned.Within 1 year after the end of treatment with NMN or placebo
  the condition of newborn births
Metabolism-related index | Within three months after the end of treatment with NMN or placebo
  Intestinal flora and metabolite changes
Metabolism-related index | Within three months after the end of treatment with NMN or placebo
  HOMA index
Metabolism-related index | Within three months after the end of treatment with NMN or placebo
  waist-hip ratio
Metabolism-related index | Within three months after the end of treatment with NMN or placebo
  BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Patients' information is requested to be confidential.